CLINICAL TRIAL: NCT01147835
Title: Effects of Herbal Lollipops on Streptococcus Mutans Levels and the Dental Caries Experience of Children With Asthma Taking beta2-adrenergic Agonist Drugs
Brief Title: Herbal Lollipops on Oral Bacterial Levels and DMFT/Dmft Scores of Children With Asthma Using Inhalers
Acronym: Lollipops
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped and not completed
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 0337-09-FB
Record Dates: First submitted 2010-06-11; First posted 2010-06-22 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Asthma; Dental Caries
Keywords: Herbal lollipops; Asthma; Dental Caries; Streptococcus mutans levels; DMFT/dmft scores
MeSH Terms: conditions — Asthma; Dental Caries | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Lollipop (Placebo Comparator): The placebo group will ingest the same herbal lollipop formula without the active ingredient.
  Interventions: Dietary Supplement: Chinese Licorice Root
- Chinese Licorice Root (Experimental): The experimental group will ingest the herbal lollipop formula with the active ingredient.
  Interventions: Dietary Supplement: Chinese Licorice Root

INTERVENTIONS:
Dietary Supplement: Chinese Licorice Root — Chinese Licorice Root lollipops are given to the subjects in the study group to ingest twice daily for 10 days. Then the subjects must wait 3 months, and then again ingest the lollipops twice daily for 10 days.
  Other Names: Herbal lollipops, Glycyrrhiza uralensis

SUMMARY:
Young children with asthma who use drugs for their asthma are at higher risk for tooth decay. These drugs can cause (1) dry mouth from less saliva secretion and (2) acid mouth that causes teeth to become soft and bacteria to multiply. Herbal lollipops may reduce the risks of tooth decay in young children. The purpose of this research is to determine how well herbal lollipops can improve the negative effects of asthma drugs over a 6-month period. Herbal lollipops contain Chinese licorice root.

DETAILED DESCRIPTION:
This study is entitled, "Effects of herbal lollipops on Streptococcus Mutans levels and the dental caries experience of children with asthma taking beta2-adrenergic drugs." In this study, forty-five (45) children between the ages of four (4) and sixteen (16) with bronchial asthma taking a beta2-adrenergic agonist drug at least once a week will participate in a six (6) month regimen of herbal lollipops as adjunctive oral hygiene therapy. The objective of this study is to determine how effective the six-month regimen of herbal lollipops is at controlling the Streptococcus Mutans levels and the caries process in the study group. Whether or not a case can be made for including herbal lollipops in standard oral hygiene protocol for children with asthma will also be a goal of this study. Relevant data will be collected using the following method. The subjects of this study will be provided with and instructed to dissolve two (2) herbal lollipops by mouth per day for the first ten (10) days of the study and again for ten (10) days three (3) months into the study. Each subject will receive a total of forty (40) lollipops for the study. The study group will be matched with a control group of forty-five (45) children who also have asthma and who take beta2-adrenergic agonist drugs as needed for symptoms. The children in the control group will be given placebo lollipops and will be instructed to use them in the manner described above. All ninety (90) subjects will be drawn from the collective patient pools of the UNMC College of Dentistry in Lincoln, NE, and the UNMC Pediatric Dentistry and UNMC Pediatrics Clinics in Omaha, NE. Oral hygiene instructions will be given to all participating subjects at the onset of the study. Entrance Streptococcus mutans levels and decayed, missing and filled teeth scores (DMFT/dmft) will be determined on the subjects and changes over the six (6) month study will be compared and evaluated. If some stabilization or improvement in the Streptococcus mutans levels and/or dental caries experience in the study group is shown, such promising results will allow for implementation of longer-term studies. The significance of this study is that adjunctive oral hygiene therapy that employs herbal lollipops may prove to help children who suffer from bronchial asthma lower their dental caries risks and have healthier oral environments unburdened by the effects of their medication and condition.

ELIGIBILITY:
Inclusion Criteria:

* Must have a medical diagnosis of asthma and must use a beta2-adrenergic agonist inhaler or nebulizer for their symptoms as needed.
* Must not have any other serious medical conditions that require taking another illness-related medication that may cloud the study results. (i.e. medications that have been shown to have anti-sialogogue effects.
* Must not have a history of severe early childhood caries (SECC) or "baby bottle tooth decay."
* Must fall within the age range of four (4) to sixteen (16) years old.
* Must be available to return for data collection during six (6) months of participation in the experiment.

Exclusion Criteria:

* Children who do not fall within all the aforementioned inclusion criteria will not be considered for participation in this study.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-09-23 (Actual); Primary Completion 2011-09-27 (Actual); Study Completion 2011-09-27 (Actual)

PRIMARY OUTCOMES:
Levels of oral Streptococcus mutans | Measured at baseline and 6 months.
  The count of S. mutans will be obtained by culture and be expressed in colony forming units (CFUs).

SECONDARY OUTCOMES:
DMFT/dmft score changes | Measured at baseling and 6 months.
  Decayed, missing and filled teeth (DMFT/dmft) score is an index for measuring dental caries.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hamilton, DDS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Kargul B, Tanboga I, Ergeneli S, Karakoc F, Dagli E. Inhaler medicament effects on saliva and plaque pH in asthmatic children. J Clin Pediatr Dent. 1998 Winter;22(2):137-40. PMID 9643188
- [Background] Ryberg M, Moller C, Ericson T. Effect of beta 2-adrenoceptor agonists on saliva proteins and dental caries in asthmatic children. J Dent Res. 1987 Aug;66(8):1404-6. doi: 10.1177/00220345870660082401. PMID 2887602
- [Background] Ryberg M, Moller C, Ericson T. Saliva composition and caries development in asthmatic patients treated with beta 2-adrenoceptor agonists: a 4-year follow-up study. Scand J Dent Res. 1991 Jun;99(3):212-8. doi: 10.1111/j.1600-0722.1991.tb01887.x. PMID 1871531
- [Background] Reddy DK, Hegde AM, Munshi AK. Dental caries status of children with bronchial asthma. J Clin Pediatr Dent. 2003 Spring;27(3):293-5. PMID 12739694
- [Background] McDerra EJ, Pollard MA, Curzon ME. The dental status of asthmatic British school children. Pediatr Dent. 1998 Jul-Aug;20(4):281-7. PMID 9783301
- [Background] Hetzer R, Heim K, Borst HG, Amende I, Sigwart U. [Cineradiographical studies of local ventricular motility before and after aorto-coronary bypass (author's transl)]. Thoraxchir Vask Chir. 1976 Aug;24(4):296-302. doi: 10.1055/s-0028-1095932. German. PMID 1086008
- [Background] Shulman JD, Taylor SE, Nunn ME. The association between asthma and dental caries in children and adolescents: A population-based case-control study. Caries Res. 2001 Jul-Aug;35(4):240-6. doi: 10.1159/000047464. PMID 11423718
- [Background] Milano M, Lee JY, Donovan K, Chen JW. A cross-sectional study of medication-related factors and caries experience in asthmatic children. Pediatr Dent. 2006 Sep-Oct;28(5):415-9. PMID 17036706
- [Background] He J, Chen L, Heber D, Shi W, Lu QY. Antibacterial compounds from Glycyrrhiza uralensis. J Nat Prod. 2006 Jan;69(1):121-4. doi: 10.1021/np058069d. PMID 16441081